CLINICAL TRIAL: NCT00553215
Title: Bladder Cancer Prognosis Programme (Incorporating SELENIB Trial) [QOL]
Brief Title: Quality of Life in Patients With Bladder Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Birmingham (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000574081; CRUK-BCPP-2005-01-QOL; ISRCTN13889738; EU-20768
Record Dates: First submitted 2007-11-02; First posted 2007-11-05 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2010-02

CONDITIONS: Bladder Cancer
Keywords: transitional cell carcinoma of the bladder; stage 0 bladder cancer; stage I bladder cancer; stage II bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

INTERVENTIONS:
Procedure: quality-of-life assessment
Procedure: questionnaire administration

SUMMARY:
RATIONALE: Studying quality of life in patients with bladder cancer may help determine the long-term effects of bladder cancer and may help improve the quality of life for patients in the future.

PURPOSE: This clinical trial is studying quality of life in patients with bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To study the effects of recurrence and progression on health-related quality of life (HRQL).
* To study the effects of repeat cystoscopy on HRQL.
* To study the patients' assessments of a hypothetical prognostic model and how this affects their preference for the mode of surveillance.

OUTLINE: This is a multicenter study.

Quality-of-life questionnaires developed by the European Organization for Research and Treatment for Cancer (EORTC) will be used. The EORTC QLQ-BLS24 with 24 questions specific to non-muscle-invasive bladder cancer and the EORTC QLQ-BLM30 with 30 questions specific to muscle-invasive bladder cancer will be combined and used in conjunction with the general cancer questionnaire QLQ-C30.

Assessments using the QLQ-C30 will be made at baseline in the entire cohort of patients. Follow-up assessments using the QLQ-C30, QLQ-BLS24, and QLQ-BLM30 167 will be made at first routine follow-up and annually until the end of study.

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Enrolled on parent protocol CRUK-BCPP-2005-01
* Bladder lesion with cystoscopic characteristics compatible with urothelial cancer or transitional cell carcinoma meeting 1 of the following criteria:

  * Non-muscle-invasive tumor
  * Muscle-invasive tumor
  * Solitary G1 pTa tumor

Exclusion criteria:

* Previous diagnosis of cancer of the urethra, bladder, ureter, or renal pelvis within the 10 years prior to current diagnosis

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Fit for cystoscopy and surgical biopsy/resection

Exclusion criteria:

* HIV infection
* Any condition that, in the opinion of the local investigator, might interfere with the safety of the patient or evaluation of the study objectives

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2700
Dates: Start 2005-12

PRIMARY OUTCOMES:
Quality of life as measured by EORTC QLQ-C30, QLQ-BLS24, and QLQ-BLM30 questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Maurice Zeegers, MD, Study Chair — University of Birmingham
Locations (1):
- University of Birmingham, Birmingham, England, United Kingdom